CLINICAL TRIAL: NCT00321802
Title: Paroxysmal Atrial Fibrillation: Role of Inflammation, Oxidative Stress Injury and Effect of Statins
Acronym: PAFRIOSIES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Anne M. Gillis, MD, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18108
Record Dates: First submitted 2006-05-03; First posted 2006-05-04 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; statin therapy; CRP levels; Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients randomized to active drug, then AF burden and CRP values will be compared to those in placebo arm.
  Interventions: Drug: Simvastatin
- 2 (Placebo Comparator): Patients take placebo once daily for 6 Months, then AF burden and CRP values will be compared to those in experimental arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — Patients take 40 mg of simvastatin per day for 6 months.
  Other Names: Zocor
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effect of statin therapy for prevention of atrial fibrillation (AF) in pacemaker and non-pacemaker patients with paroxysmal atrial fibrillation in the absence of significant coronary artery disease.

DETAILED DESCRIPTION:
Patients with a history of paroxysmal atrial fibrillation, with or without a dual chamber pacemaker and who meet all study criteria, will be randomized to receive either a placebo, or simvastatin 40 mg, daily for 6 months.

Liver enzymes are drawn at randomization and 3 months. CRP and oxidative stress products are drawn at randomization, weekly for the first month and then monthly for 5 months.

Patients transmit their rhythm, twice daily for 5 consecutive days at randomization, then 5 consecutive days monthly for 6 months.

Clinic visits are required at randomization, 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal AF (> 3 epis each > 15 min in length) over 6 months
* Patients on stable antiarrhythmic drug therapy and life expectancy > 1 year

Exclusion Criteria:

* Patients with PAF due to reversible cause
* Chronic inflammatory conditions
* Other medical conditions requiring statin therapy
* Patients on amiodarone or verapamil
* Elevated CK or ALT
* Life expectancy <1 year
* TAVN ablation
* Geographic isolation
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Time to first detected AF | 6 Months

SECONDARY OUTCOMES:
Changes in CRP and oxidative stress levels over time and their relationship with AF burden | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Gillis, MD, Principal Investigator — University of Calgary; Henry J Duff, MD, Study Director — University of Calgary; Derek V Exner, MD, MPH, Study Director — University of Calgary; Katherine Kavanagh, MD, Study Director — University of Calgary; L B Mitchell, MD, Study Director — University of Calgary; Robert S Sheldon, MD, PhD, Study Director — University of Calgary; D G Wyse, MD, PhD, Study Director — University of Calgary; George Veenhuyzen, MD, Study Director — University of Calgary
Locations (1):
- University of Calgary, Foothills Hospital, Calgary, Alberta, Canada